CLINICAL TRIAL: NCT01246934
Title: Segment Transport Versus Acute Shortening In The Treatment of Tibial Pseudarthroses With Bone Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BVUORT001
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: TIBIA PSEUDOARTHROSES

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- COMPLICATION (No Intervention)
  Interventions: Other: ASR METHOD

INTERVENTIONS:
Other: ASR METHOD

SUMMARY:
In this study the investigators are presenting the advantages as well as the disadvantages of ACUTE SHORTENING AND RELENGTHENINIG VS SEGMENT TRANSPORT methods.

ELIGIBILITY:
Inclusion Criteria:TIBIA PSEUDOARTHROSES -

Exclusion Criteria:BONE LOSS GREATER THAN 10 CM

-

Ages: 13 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
TREATMENT PERIOD AND COMPLICATION RATE

CONTACTS AND LOCATIONS:
Locations (1):
- Cengiz Sen, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Paley D, Sen C, Tetsworth K. Acute Shortening With Subsequent Relengthening Versus Bone Transport In The Treatment Of Tibial Bone Defect, 11th Asami North America Annual Scientific Meeting, February 18-25, Berkeley Ca, 2001